CLINICAL TRIAL: NCT05235620
Title: An Evaluation of the Spread and Scale of PatientToc™ From Primary Care to Community Pharmacy Practice for the Collection of Patient-Reported Outcomes: Phase 2
Brief Title: Evaluation of PatientToc in Community Pharmacies
Status: Enrolling by invitation | Type: Observational
Sponsor: Purdue University (Other)
Collaborators: University of Wisconsin, Madison (Other); University of Minnesota (Other); University of Arkansas (Other); L.A. Net Community Health Resource Network (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Indiana Clinical and Translational Sciences Institute (Other)
Responsible Party: Principal Investigator, Margie Snyder, Associate Professor of Pharmacy Practice, Purdue University
Other Study IDs: 2008163459
Record Dates: First submitted 2022-01-11; First posted 2022-02-11 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence | interventions — Pharmacies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pharmacy staff: Pharmacy staff working at pharmacies which have chosen to implement PatientToc software for this implementation science project and evaluation. Pharmacy staff will be observed and participate in interviews pertaining to their experiences using PatientToc.
  Interventions: Other: PatientToc use in pharmacies
- Pharmacy patients: Patients engaged in completing medication adherence-related questionnaires in the PatientToc software at their pharmacies. Patient-level medication, health history, and self-reported adherence information will be collected from patients meeting eligibility criteria. Patients will also be observed and interviewed about their experiences using PatientToc.
  Interventions: Other: PatientToc use in pharmacies

INTERVENTIONS:
Other: PatientToc use in pharmacies — PatientToc has been adapted for use in pharmacies. Patients using specific medications will be prompted to complete questionnaires about their self-reported adherence.

SUMMARY:
The purpose of this study is to evaluate the initial "spread and scale" of PatientToc™, a patient-reported outcomes (PROs) collection software, to community pharmacies for the collection and use of PROs data pertaining to medication adherence. The investigators are doing this by engaging PatientToc™ and pharmacy partners in two plan-do-study-act (PDSA) cycles to implement and refine PatientToc™ and an implementation toolkit (i.e., supports/resource tools) within a small number of community pharmacies. Investigators will then scale implementation to more community pharmacies in a rigorous theory-driven evaluation of PatientToc™ implementation using interviews, self-reported data from the pharmacy, observations, and administrative data. Collectively, the findings will inform long-term collection and use of PROs data pertaining to medication use.

DETAILED DESCRIPTION:
Medication non-adherence is a problem of critical importance, affecting approximately 50% of all persons taking at least one regularly scheduled prescription medication and costing the United States more than $100 billion annually. Medication non-adherence is associated with clinical outcomes including hospitalizations and mortality. It is a complex, multi-faceted problem with many causes such as forgetfulness, access/affordability concerns, and avoiding medication due to bothersome side effects. Johnson's Medication Adherence Model (MAM) summarizes these causes by theorizing that patients must both "Remember" and "Intend" to take medication. The importance of reducing medication non-adherence is reflected in the Healthy People 2020 goals and objectives and recognized in the Centers for Medicare and Medicaid Services (CMS) star ratings program for Medicare Part D prescription drug plans (PDPs). Plans are rated annually as achieving 1 (lowest quality) to 5 (highest quality) stars. Plans receiving 5 stars are rewarded through quality bonus payments and the ability for patients to switch to the plan outside of the annual open enrollment period. Several measures used in determining star ratings are based on beneficiary medication adherence.

Community pharmacists are uniquely positioned to intervene on medication non-adherence. Community pharmacies are widely accessible and visited frequently by patients with chronic conditions, including the elderly and patients without a regular source of primary care. Community pharmacists can provide support for challenges commonly faced by patients such as limited health literacy, being un/underinsured, and limited English proficiency. Further, community pharmacies nationwide have increased efforts to improve measures influencing PDP star measures to ensure the pharmacy is positioned for financial reward through inclusion in the PDPs preferred pharmacy network and possible bonus payments. Traditional data sources for identifying and resolving medication non-adherence in community pharmacies include prescription fill histories. However, medication possession does not necessarily mean patients are taking medications as prescribed. Patient-reported outcomes (PROs), measuring adherence challenges pertaining to both remembering and intention to take medication, offer a rich data source for pharmacists and prescribers to use to resolve medication non-adherence.

Although the value of collecting and utilizing PROs for clinical and research purposes has been more widely recognized in recent years, to the investigators' knowledge, there are no examples of widespread electronic collection and use of PROs data 1) in community pharmacy settings, or 2) pertaining specifically to medication adherence in ambulatory settings. Moreover, numerous implementation challenges have been reported and the systematic collection of timely and actionable PROs data can be challenging, particularly for patient populations with limited literacy and/or health literacy. For example, paper-based data collection can be burdensome for data management/analysis and data quality concerns may be evident. Electronic data collection offers advantages but technology must ensure privacy and security standards are in place to support the reliability and validity of the data. In addition, data must be accessible to providers in a timely fashion for clinical decision making. Finally, while technology exists to facilitate the transfer of PROs data into electronic health records (EHRs) and providers want these data to populate with laboratory results, few electronic systems do so.

In December 2016, the Agency for Healthcare Research and Quality (AHRQ) released Funding Opportunity Announcement PA-17-077 which provides funding for research projects to "scale and spread" successful health information technology models that use PROs in ambulatory settings. Consequently, the investigators received funding in April 2019 to conduct research to inform long-term collection and use of PROs data pertaining to medication adherence in community pharmacies by spreading and scaling a successful model (PatientToc™, described below) for health information technology-enabled PROs collection.

Description of PatientToc: Current Use in Physician Offices PatientToc™ is a PROs collection software developed by investigators from the L.A. Net Community Health Resources Network (LA Net), a primary care practice-based research network (PBRN) in California. PatientToc™ was developed to facilitate collection of PROs data from low-literacy and non-English speaking patients in Los Angeles. L.A. Net provided a design for the product based on experience collecting PROs from more than 10,000 patients in L.A. Net practices speaking 42 different languages. The system was developed over a period of 4 years with continuous input from clinicians, community health workers, patients and researchers. PatientToc™ is used in waiting rooms, pre-visit areas, exam rooms, and educator rooms. Patients interact with a 10-inch android tablet that is either hand held or installed in a case or holder attached to a table. Consistent with research on low-literacy, the system presents one question at a time. Patients use disposable ear buds to maintain confidentiality when patients use the read aloud function. The system can deliver any PROs and responses are transmitted real time to the PatientToc™ server where staff and clinicians can access the results both as a pdf replica of a paper version of the completed survey, and as an aggregated SQL or Excel database. PatientToc™ integrates with EHRs via Health Level Seven (HL7) standards or Fast Healthcare Interoperability Resources (FHIR) interfaces, and through third party integration with service provider systems. Currently, PatientToc™ is being used in over 36 practices including 2 Federally Qualified Health Centers. Two California health plans have also used the system to transmit mandatory initial health assessments. Approximately 10,000 patients have completed PROs on PatientToc™ tablets, including the: PHQ-9, Medicare Health Risk Assessments, SBIRT screening, and others.

Aim 1: Conduct a pre-implementation developmental formative evaluation to determine community pharmacy workflow and current practices for identifying and resolving medication non-adherence, potential barriers and facilitators to PatientToc™ implementation, and create a draft implementation toolkit. This Aim was previously completed under a separate exempt protocol

Aim 2: Conduct two plan-do-study-act (PDSA) cycles to refine an implementation toolkit for spreading and scaling implementation of PatientToc™ in community pharmacies.

Aim 3: Conduct a comprehensive, theory-driven evaluation of the quality of care, implementation, and patient health outcomes of spreading and scaling PatientToc™ to community pharmacies.

Aim 4: To explore the feasibility of linking PROs data from PatientToc™ with healthcare utilization data. This will inform future research.

Aim 5: To conduct exploratory and secondary analyses to examine variations in medication therapy problems (MTPs), pharmacist interventions, and PatientToc™ outcomes by implementation scope and patient characteristics. Secondary analyses using Aim 1 data might also be completed, such as examining expected barriers from a staff perspective vs. actual concerns identified in Aims 2 and 3 pertaining to feasibility and acceptability.

Aim 6: To evaluate a novel continuing education (CE) program provided to pharmacies as part of the PatientToc™ implementation toolkit.

Aim 7: To assess participating pharmacists' perceptions of participating in this study.

ELIGIBILITY:
Pharmacist/pharmacy staff eligibility criteria:

* Aged 18 years or older
* Employee (paid) or PharmD rotation student trainee/volunteer at the pharmacy during the time of PatientToc™ implementation

Pharmacy patient eligibility criteria:

The specific pharmacy workflow for introducing patients to PatientToc™ may vary by participating pharmacy. For example, all pharmacy patients might have the opportunity to complete PROs in the tablet/mobile application (if desired by the pharmacy) with only a subset included in our evaluation. This variation does not change our study/evaluation procedures and is allowed to facilitate successful PatientToc™ implementation in patient care.

For the purposes of this evaluation, individual-level data will be sought from patients who are:

* ≥ 50 years of age
* Have one or more specific chronic conditions (i.e., hypertension, Type 2 diabetes, and dyslipidemia; per self-report, ICD code if available, and/or inferred by medications filled) requiring routine (regularly scheduled, not "as needed" dosing)
* Medications are oral (solid dosage form)
* Prescription medication filled at least once previously by the study pharmacy as 30-day supplies. In situations where patients with 30-day supplies also fill some medications as 90-day (or other quantity) supplies, they will be enrolled if their first medication chosen for PROs completion was a 30-day supply.
* Baseline non-adherence as determined by responses to the BMQ PRO for one or more targeted medications, specifically, the first medication chosen for PROs completion by the patient for their primary condition of interest (hypertension, Type 2 diabetes, and dyslipidemia) when they have more than one of these conditions and take more than one targeted medication.
* Able to provide consent and read and/or comprehend English or another language for which the intervention and study materials (e.g., consent documents) is available OR has a legal representative (self-reported) with authority to act on their behalf to complete PROs/interview/other data collection and consent documents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pharmacy staff and patients at pharmacies agreeing to implement PatientToc as part of this implementation science project.
Sampling Method: Non-Probability Sample
Enrollment: 1175 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Estimated)

PRIMARY OUTCOMES:
Self-reported medication adherence, measured by Brief Medication Questionnaire | Monthly, up to 7 months
  Validated survey consisting of 4 items asking respondents to consider their medication adherence for each regularly scheduled prescription medication of interest over the past 7 days

SECONDARY OUTCOMES:
Self-reported medication adherence measured by the Merck Medication Adherence Estimator (Adherence Estimator), | Monthly, up to 7 months
  Validated 3 item questionnaire measuring self-reported adherence barriers pertaining to cost, concerns, and commitment for specific medications
Medication regimen complexity measured by the Medication Regimen Complexity Index (MRCI), | Monthly, up to 7 months in select patients only
  Automated 65-item tool measuring regimen complexity across three components: form/route, dosing frequency, and special instructions using the patient's prescription fill data at the pharmacy
Pharmacy-level population medication adherence measured by from pharmacy-level EQuIPP data | Prior to and at the end of the intervention
  Program administered by Pharmacy Quality Solutions, Inc., that provides community pharmacies with report cards for their performance on proportion prescriptions filled for pertaining to medication use within categories of interest
Acceptability of intervention | Monthly, up to 7 months
  Perceptions among stakeholders regarding satisfaction with PatientToc implementation, as measured by qualitative themes identified through direct observation and interviews as well as descriptive statistics on refusal data (patients declining participation, skipping items)
Adoption of intervention | Monthly, up to 7 months
  The initial decision to utilize PatientToc in pharmacy practice, as measured by qualitative themes identified through direct observation and interviews as well as descriptive statistics on patient utilization (number of patients consented, measures completed)
Appropriateness of intervention | First month of implementation
  Perceived relevance and compatibility of PatientToc for community pharmacies, as measured by qualitative themes identified through direct observation and interviews.
Costs of intervention | Monthly, up to 7 months
  Descriptive statistics (mean, SD, total) of costs of implementing PatientToc at participating pharmacies.
Feasibility of intervention | Monthly, up to 7 months
  The extent to which PatientToc can be successfully used in community pharmacies, measured using a mixed methods approach combining qualitative themes identified through direct observation and interviews and number of contacts made with pharmacy to discuss issues with the intervention.
Fidelity of intervention | Monthly, up to 7 months
  The degree to which PatientToc was implemented as intended, as measured by qualitative themes identified through direct observation and interviews as well as descriptive statistics on pharmacy adherence to PatientToc implementation as directed per implementation toolkit (e.g., number of days per PDSA when PatientToc was accessed; proportion of patients for whom PatientToc data was reviewed and used by the pharmacist during (as opposed to after) patient visit to pharmacy.)
Penetration of intervention | monthly, up to 7 months
  Integration of PatientToc within community pharmacies measured by descriptive statistics on pharmacy-level utilization of PatientToc (e.g., percent of pharmacist shifts)
Sustainability of intervention | monthly, up to 7 months
  Extent to which PatientToc is maintained within community pharmacies measured by number of consecutive months goal level of patient participation achieved
Prescription transfers | monthly, up to 7 months
  Prescription transfers in and out of pharmacy (self-report) during observation period.
Prescription volume | monthly, up to 7 months
  Prescriptions dispensed by pharmacy (self-report) during observation period.
Patient satisfaction | monthly, up to 7 months
  Patient satisfaction with pharmacy services (self-report) during observation period. Items will be analyzed individually. These items will not be tabulated to create a scale.

CONTACTS AND LOCATIONS:
Overall Officials: Margie E Snyder, PharmD, MPH, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No